CLINICAL TRIAL: NCT00599833
Title: Locally Advanced Pancreatic Cancer: Phase II Study of Cetuximab and 3-D Conformal Image Guided Radiotherapy (PACER)
Brief Title: Cetuximab and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CHNT-PACER; CDR0000582420 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2006-001742-13; EU-207103; CTA-21266/0210/001-0001
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Radiotherapy, Conformal

INTERVENTIONS:
Biological: cetuximab
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving cetuximab together with 3-dimensional conformal radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with radiation therapy works in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the progression free survival rate in patients treated with cetuximab and radiotherapy.

Secondary

* To determine the response rate, toxicity of the combined regimen, and clinical benefit response in patients treated with cetuximab and radiotherapy.

OUTLINE: Patients receive cetuximab IV over 1-2 hours once weekly for 6-7 weeks. Patients also undergo concurrent 3-dimensional image-guided conformal radiotherapy in 28-30 fractions over approximately 5.5-6 weeks (2-4 hours after administration of cetuximab).

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically or cytologically confirmed diagnosis of inoperable, non-metastatic, locally advanced pancreatic adenocarcinoma
* No neuroendocrine tumors or lymphoma of the pancreas
* No extensive disease unable to be covered in a radically treatable radiotherapy volume

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* Hemoglobin ≥ 10g/dL
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³ (prior transfusions for patients with low hemoglobin allowed)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Serum urea ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Adequate biliary drainage with no evidence of active uncontrolled infection (patients on prophylactic antibiotics are eligible)
* Not pregnant or nursing
* Negative pregnancy test
* Women and men of child-bearing potential should be using an adequate contraception method, which must be continued for 3 months after completion of therapy
* No unresolved biliary tract obstruction
* No history of prior malignancy that may interfere with the response evaluation except for any of the following:

  * Cervical carcinoma in-situ treated by cone-biopsy/resection
  * Nonmetastatic basal and/or squamous cell carcinomas of the skin
  * Any early stage (stage I) malignancy adequately resected for cure greater than 5 years previously
* No relative contraindication to radiotherapy
* No evidence of severe uncontrolled systemic diseases or laboratory finding that in the view of investigator makes it undesirable for the patient to participate in the trial
* No disorder likely to impact compliance with the protocol

PRIOR CONCURRENT THERAPY:

* Must be completely recovered from previous surgery
* The following prior interventions are allowed:

  * Non-curative operation (i.e., R2 resection with macroscopic residual disease evident on CT scan or palliative bypass procedure)
  * Stent insertion in the common bile duct
* No previous radiotherapy within current treatment field
* No previous administration of EGF monoclonal antibodies, EGFR signal transduction inhibitors or EGFR-targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months

SECONDARY OUTCOMES:
Response rate by RECIST criteria
Toxicity by NCI CTCAE criteria
Clinical benefit response

CONTACTS AND LOCATIONS:
Overall Officials: Pat Price, MD, Study Chair — The Christie NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Cookridge Hospital, Leeds, England
  - Christie Hospital, Manchester, England